CLINICAL TRIAL: NCT04420962
Title: Quantifying Microbial Keratitis to Predict Outcomes
Brief Title: Automated Quantitative Ulcer Analysis Study
Acronym: AQUA
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Maria Woodward, Assistant Professor, University of Michigan
Other Study IDs: HUM00174923; R01EY031033 (NIH)
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Keratitis
Keywords: Corneal Ulcer
MeSH Terms: conditions — Keratitis; Corneal Ulcer | interventions — Visual Acuity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Microbial Keratitis: Presence of a bacteria or fungal keratitis with ≥ 2mm stromal infiltrate
  Interventions: Diagnostic Test: Visual Acuity
- Viral or Inflammatory Keratitis: Non-infectious inflammatory, Viral, Acanthamoeba, or other forms of keratitis
  Interventions: Diagnostic Test: Visual Acuity

INTERVENTIONS:
Diagnostic Test: Visual Acuity — Best corrected visual acuity utilizing the Snellen method

SUMMARY:
This is a multiple site observational study that will review patient features (clinical and morphologic) over a 90 day period during care of participants with microbial keratitis with presence of clinically significant ≥2mm stromal infiltrate compared with participants with other forms of keratitis.

DETAILED DESCRIPTION:
The primary objective of this study is to determine associations between participant features (clinical and morphologic) and best corrected visual acuity at Day 90. Imaging, focused on slit lamp photography and supplemented by other imaging markers will be collected for review. A medical record review at one year following participants initial visit will record any corneal procedure and visual acuity testing that occurred during this window. Participants will complete demographic, clinical, and standardized health surveys.

ELIGIBILITY:
Inclusion Criteria:

* Cases- microbial keratitis (bacterial or fungal) with presence of clinically significant ≥2mm stromal infiltrate
* Controls- Inflammatory, viral, Acanthamoeba, or other keratitis

Exclusion Criteria:

* Pregnancy
* Prior incisional corneal surgery
* No light perception vision
* Corneal perforation or impending perforation
* Inpatient status
* Institutional status
* Cognitively impaired
* Prisoner

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subject population will be those that seek care at an ophthalmology clinic for microbial, non-infectious, viral, Acanthamoeba, or other keratitis and agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 90 day follow up
  Visual Acuity

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Woodward, MD, MS, Principal Investigator — University of Michigan
Locations (2):
- University of Michigan- Kellogg Eye Center, Ann Arbor, Michigan, United States
- Aravind Eye Care System, Madurai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel TP, Prajna NV, Farsiu S, Valikodath NG, Niziol LM, Dudeja L, Kim KH, Woodward MA. Novel Image-Based Analysis for Reduction of Clinician-Dependent Variability in Measurement of the Corneal Ulcer Size. Cornea. 2018 Mar;37(3):331-339. doi: 10.1097/ICO.0000000000001488. PMID 29256985
- [Background] Maganti N, Tan H, Niziol LM, Amin S, Hou A, Singh K, Ballouz D, Woodward MA. Natural Language Processing to Quantify Microbial Keratitis Measurements. Ophthalmology. 2019 Dec;126(12):1722-1724. doi: 10.1016/j.ophtha.2019.06.003. Epub 2019 Jun 11. PMID 31307829
- [Background] Kriegel MF, Huang J, Ashfaq HA, Niziol LM, Preethi M, Tan H, Tuohy MM, Patel TP, Prajna V, Woodward MA. Algorithm Variability in Quantification of Epithelial Defect Size in Microbial Keratitis Images. Cornea. 2020 May;39(5):628-633. doi: 10.1097/ICO.0000000000002258. PMID 31977729
- [Background] Loo J, Kriegel MF, Tuohy MM, Kim KH, Prajna V, Woodward MA, Farsiu S. Open-Source Automatic Segmentation of Ocular Structures and Biomarkers of Microbial Keratitis on Slit-Lamp Photography Images Using Deep Learning. IEEE J Biomed Health Inform. 2021 Jan;25(1):88-99. doi: 10.1109/JBHI.2020.2983549. Epub 2021 Jan 5. PMID 32248131
- [Background] Lu MC, Deng C, Greenwald MF, Farsiu S, Prajna NV, Nallasamy N, Pawar M, Hart JN, Sr S, Kochar P, Selvaraj S, Levine H, Amescua G, Sepulveda-Beltran PA, Niziol LM, Woodward MA; and the AQUA Study Team. Automatic Classification of Slit-Lamp Photographs by Imaging Illumination. Cornea. 2024 Apr 1;43(4):419-424. doi: 10.1097/ICO.0000000000003318. Epub 2023 May 31. PMID 37267474
- [Background] Woodward MA, Vogt EL, Niziol LM, Mian SI, Sugar A, Verkade A, Nallasamy N, Pawar M, Kang L, Miller KD, Winter S, Farsiu S, Prajna NV. Factors Associated with Vision Outcomes in Microbial Keratitis: A Multisite Prospective Cohort Study. Ophthalmology. 2025 Jul;132(7):830-841. doi: 10.1016/j.ophtha.2025.02.004. Epub 2025 Feb 8. PMID 39929390
- [Derived] Vogt EL, Niziol LM, Yang Z, Wang Y, Pawar M, Dmitriev P, Gupta AS, Armenti ST, Hood CT, Shtein RM, Kipley MM, Lee MC, Sumithra SR, Thulukanam M, Kochar P, Selvaraj S, Redd TK, Prajna NV, Farsiu S, Woodward MA. Association of Deep Learning Imaging Algorithm Measures of Microbial Keratitis With Vision Outcomes. Cornea. 2025 Oct 29. doi: 10.1097/ICO.0000000000004029. Online ahead of print. PMID 41247284
- [Derived] Lee MC, Vogt EL, Hicks PM, Pawar M, Lu MC, Niziol LM, Terek DA, Nallasamy N, Hakim FE, Woodward MA. Social Risk Factors Associated With Microbial Keratitis. Cornea. 2026 Jan 1;45(1):21-28. doi: 10.1097/ICO.0000000000003766. Epub 2024 Dec 10. PMID 39661074